CLINICAL TRIAL: NCT00143338
Title: A Phase 2, Exploratory Study to Examine the Effects of Inhaled Insulin, Compared With Subcutaneously Administered Insulin, on Airway Lining Fluid Composition in Subjects With Type 2 Diabetes Mellitus.
Brief Title: To Examine the Lung When People With Diabetes Take an Inhaled Form of Insulin, Compared to Subcutaneous Insulin.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A2171053
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2008-02-12 (Estimated); Status verified 2008-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

INTERVENTIONS:
Drug: Inhaled insulin

SUMMARY:
To examine the lung when people with diabetes take an inhaled form of insulin, compared to subcutaneous insulin.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes Mellitus
* Normal lung function

Exclusion Criteria:

* Smokers

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20
Dates: Start 2004-11; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
To assess in patients with type 2 diabetes mellitus the effects, if any, on lung lining fluid cell count and differential within subjects after 12 weeks of inhaled insulin therapy compared to 12 weeks of subcutaneous short-acting therapy.

SECONDARY OUTCOMES:
(1) Albumin and fibrinogen concentrations, and airway appearance in the above subjects. (2) routine safety, tolerance, and efficacy in the above subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Pfizer Investigational Site, Fresno, California
  - Pfizer Investigational Site, San Antonio, Texas

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A2171053&StudyName=To+Examine+the+Lung+When+People+with+Diabetes+Take+an+Inhaled+Form+of+Insulin%2C+Compared+to+Subcutaneous+Insulin%2E